CLINICAL TRIAL: NCT04217486
Title: Will Visual Affirmation of Knee Range of Motion (ROM) Affect Patient Outcomes in Patients Undergoing a Primary Total Knee Arthroplasty (TKA)? A Prospective, Randomized Study.
Brief Title: ROM Outcomes in Patients Undergoing a Primary TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Arthur Malkani, Professor, Adult Reconstruction, Dept. of Orthopaedic Surgery, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19.1179
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Postoperative Period

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - will be shown their photograph at 2 weeks post-operative. (Experimental): 40-50 arms: patients undergoing a unilateral, cementless primary TKA, secondary to osteoarthritis will be shown a photograph of their knee, photographed in maximum flexion and extension, at 2 weeks postoperatively.
  Interventions: Other: Patient will be shown a photograph of their knee at 2 weeks postop
- B - will not be shown their photograph (Active Comparator): 40-50 arms: patients undergoing a unilateral, cementless primary TKA, secondary to osteoarthritis will not be shown a photograph of their knee, photographed in maximum flexion and extension, at 2 weeks postoperatively.
  Interventions: Other: Patient will not be shown a photograph of their knee at 2 weeks postop

INTERVENTIONS:
Other: Patient will be shown a photograph of their knee at 2 weeks postop — Patients who undergo primary TKA surgery will then be shown a photograph of their knee at 2 weeks postoperative.
  Arms: A - will be shown their photograph at 2 weeks post-operative.
Other: Patient will not be shown a photograph of their knee at 2 weeks postop — Patients who undergo primary TKA surgery will not be shown a photograph of their knee at 2 weeks postoperative.
  Arms: B - will not be shown their photograph

SUMMARY:
The goal of this prospective, randomized study is to compare the outcomes of patients undergoing primary TKA after photographing final knee range of motion immediately post-operatively and sharing these photographs with patients at their first follow-up appointment versus a group that does not see a photograph.

DETAILED DESCRIPTION:
The goal of this prospective, randomized study is to compare the outcomes of patients undergoing primary total knee arthroplasty (TKA) after photographing final knee range of motion immediately postoperatively and sharing these photographs with patients at their first follow-up appointment versus a group that does not see a photograph. The knee will be photographed in maximum flexion and extension. The primary objectives will be to compare the range of motion of the operative knee at 2 weeks and 6 weeks postoperatively. In the investigator's institution, patients who have failed to achieve 90 degrees of flexion at a postoperative period of 6 weeks undergo manipulation of the knee under anesthesia (MUA). The investigators will also measure how many patients require MUA in the photograph group and non-photograph group. MUA will be performed if patients fail to achieve 90 degrees of flexion at 6 weeks post-op.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between the age of 22-89
2. Patient is scheduled to undergo a unilateral, cementless primary TKA, secondary to osteoarthritis
3. Patient agrees to participate as a study subject and signs the Informed Consent and Research Authorization documents
4. Patient is able to read and speak English.

Exclusion Criteria:

1. Patient is under the age of 22 or over the age of 89
2. Patient has preoperative stiffness/contracture of the knee secondary to post-traumatic arthritis
3. Patient is scheduled to undergo a bilateral TKA surgery
4. Patient is unable to read and speak English

Ages: 22 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
total length of hospital stay | outcome measure will be taken at 2 weeks postoperatively
  total length of hospital stay as defined by number of days from date of surgery to date of discharge
Knee Society Score | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery)
  Knee Society Score. The score is on a scale from 0-100. A higher value represents a better outcome.
Knee Society Score | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Knee Society Score. The score is on a scale from 0-100. A higher value represents a better outcome.
WOMAC Score | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery)
  WOMAC score. The score is on a scale from 0-100. In contrast to the Knee Society Score, on the WOMAC a lower value represents a better outcome
WOMAC Score | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  WOMAC score. The score is on a scale from 0-100. In contrast to the Knee Society Score, on the WOMAC a lower value represents a better outcome
Active range-of-motion (ROM) | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery)
  Active ROM (range-of-motion) as measured by a goniometer (range of 0-135 degrees)
Active range-of-motion (ROM) | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Active ROM (range-of-motion) as measured by a goniometer (range of 0-135 degrees)
Incidence of loss of knee motion requiring an MUA (manipulation under anesthesia) | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Loss of knee motion is defined as failure to achieve greater than 100 degrees of active flexion. Manipulation under anesthesia is an outpatient procedure performed by orthopedic surgeon to help improve patient's range-of-motion.
Operative Time | outcome measure will be taken at 2 weeks postoperatively
  Total Operative Time as defined in minutes
Tourniquet time | outcome measure will be taken at 2 weeks postoperatively
  Total Tourniquet Time is the number of minutes that the tourniquet is inflated, as defined in minutes.
Estimated Blood Loss (EBL) | outcome measure will be taken at 2 weeks postoperatively
  Estimated Blood Loss as defined by the amount of intraoperative blood loss measured in cubic centimeters (cc).

SECONDARY OUTCOMES:
Number of Participants with postoperative complications | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Number of Participants with postoperative complications. A postoperative complication is defined as any diagnosis or condition that necessitates a re-operation or procedure on the surgical knee

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Malkani, MD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No